CLINICAL TRIAL: NCT03897205
Title: A Randomized, Open-Label, Multi-Centre, Active Control, Efficacy and Safety Study of Imlifidase in Eliminating Donor Specific Anti-HLA Antibodies in the Treatment of Active Antibody-Mediated Rejection in Kidney Transplant Patients
Brief Title: An Efficacy and Safety Study of Imlifidase in Treatment of Antibody-Mediated Rejection in Kidney Transplant Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hansa Biopharma AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-HMedIdeS-12; 2018-000022-66 (EudraCT Number)
Record Dates: First submitted 2019-03-27; First posted 2019-04-01 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Kidney Transplant Rejection
MeSH Terms: interventions — Mac-1-like protein, Streptococcus; Plasma Exchange

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Imlifidase (Experimental): Subjects randomized to imlifidase treatment received one intravenous dose of imlifidase, 0.25 mg/kg, administered over 15 minutes.
  Interventions: Drug: Imlifidase
- Plasma Exchange (Active Comparator): Subjects randomized to plasma exchange (PE) treatment received 5-10 sessions of PE, as judged by the investigator. Immunoadsorption (IA) could replace PE, at the discretion of the investigator.
  Interventions: Other: Plasma Exchange

INTERVENTIONS:
Drug: Imlifidase — Imlifidase is an immunoglobulin G (IgG) degrading enzyme of Streptococcus pyrogenes that cleaves all 4 human subclasses of IgG with strict specificity.
  Other Names: HMED-IdeS, IdeS, IgG endopeptidase
  Arms: Imlifidase
Other: Plasma Exchange — The subject's plasma is removed and discarded and the subject receives replacement donor plasma, albumin, or a combination of albumin and saline. IA may be used instead of PE to the discretion of the investigator. IA is achieved by passing a subject's plasma over columns that bind immunoglobulins and then the plasma is passed back to the subject.
  Arms: Plasma Exchange

SUMMARY:
The purpose of this study was to investigate how efficiently the study medication imlifidase reduces the amount of donor specific antibodies (DSA) in comparison with plasma exchange (PE) therapy, in patients who have had an active or chronic active antibody mediated rejection (AMR) after being kidney transplanted. The purpose was also to investigate and compare safety for these two treatments.

DETAILED DESCRIPTION:
Antibodies to human leukocyte antigens (HLAs) have a strong correlation with allograft injury and loss. Treatment with imlifidase, PE and immunoabsorption (IA) all aim to reduce antibody levels.

This study compared the reduction in DSA levels after treatment with imlifidase and PE in patients diagnosed with active or chronic active AMR (according to Banff 2017 or Banff 2019 criteria) having at least a 25% rise in serum creatinine compared with last measurement prior to the AMR. (Patients with delayed graft function and AMR within 10 days after kidney transplantation could be included regardless of serum creatinine level.) Eligible patients were randomized to either 1 dose of imlifidase (0.25 mg/kg) or 5-10 sessions of PEs (IA could replace PE at the discretion of the investigator).

All patients received pulse methylprednisolone Day 1 to Day 3, followed by a tapering schedule with prednisolone/prednisone. Patients randomised to imlifidase received their first dose of methylprednisolone before imlifidase was administered. The patients did also receive high dose intravenous immunoglobulin (IVIg) 3 days after imlifidase treatment or directly after the last PE. In addition a single dose of rituximab was given 5 days after completed IVIg infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent obtained before any study-related procedures
2. Willingness and ability to comply with the protocol
3. Male and/or female donor kidney recipients age ≥18 years at the time of screening
4. Presence of DSA(s)
5. Meet the Banff 2017 criteria for active or chronic active AMR
6. At least 25% rise in serum creatinine compared to last individual value taken prior to the AMR. Patients with delayed graft function and AMR within 10 days after transplant (confirmed by kidney biopsy) can be included regardless of serum creatinine level
7. Women of child-bearing potential willing or able to use at least one highly effective contraceptive method throughout the study. In the context of this study, an effective method is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly
8. Men willing to use double-barrier contraception from the first day of treatment until at least 2 months after the dose of imlifidase, if not abstinent

Exclusion Criteria:

1. Previous treatment with imlifidase
2. Previous high dose IVIg treatment (2 g/kg) within 28 days prior to inclusion
3. Lactating or pregnant females
4. Significantly abnormal general serum screening lab results judged inappropriate for inclusion in the study by the investigator
5. Intake of other investigational drugs within 5 half-lives (or similar) of the product prior to inclusion
6. Clinically relevant active infection(s) as judged by the investigator
7. Any condition that in the opinion of the investigator could increase the subject's risk by participating in the study such as severe immune deficiency and severe cardiac insufficiency [New York Heart Association (NYHA) Class IV] or severe uncontrolled heart disease
8. Known allergy/sensitivity to imlifidase, IVIg and/or rituximab and the respective excipients
9. Patient unable to tolerate treatment with plasmapheresis or immunoadsorption, as judged by the investigator
10. Unsuitable to participate in the study for any other reason as judged by the investigator
11. Positive polymerase chain reaction (PCR) test for severe acute respiratory syndrome corona virus 2 (SARS-CoV-2) infection
12. Current diagnosis or history of thrombotic thrombocytopenic purpura (TTP), or known familial history of TTP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2022-05-28 (Actual); Study Completion 2022-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Operations, Study Director — Hansa Biopharma AB
Locations (14):
- United States (4):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Brigham and Women Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - New York University Grossman School of Medicine, New York, New York
- Australia (3):
  - The Royal Melbourne Hospital, Melbourne, Victoria
  - Royal Adelaide Hospital, Adelaide
  - Royal Prince Alfred Hospital, Sydney
- Universitätsklinik für Innere Medizin III, Klinische Abteilung für Nephrologie MUW, Vienna, Austria
- France (4):
  - Hôpital Pellegrin, Bordeaux
  - CHU Grenoble Alpes - Néphrologie, dialyse et transplantation, Grenoble
  - Hôpital Saint-Louis. Service de Néphrologie et Transplantation, Paris
  - Hôpital Necker - Service de Néphrologie - Transplantation, Paris
- Germany (2):
  - Charité-Universitätsmedizin. Dept. of Nephrology and Medical Intensive Care, Berlin
  - Medizinische Hochschule Hannover, Hanover

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Halleck F, Bohmig GA, Couzi L, Rostaing L, Einecke G, Lefaucheur C, Legendre C, Montgomery R, Hughes P, Chandraker A, Wyburn K, Halloran P, Maldonado AQ, Sjoholm K, Runstrom A, Lefevre P, Tollemar J, Jordan S. A Randomized Trial Comparing Imlifidase to Plasmapheresis in Kidney Transplant Recipients With Antibody-Mediated Rejection. Clin Transplant. 2024 Jul;38(7):e15383. doi: 10.1111/ctr.15383. PMID 39023092

RESULTS

PARTICIPANT FLOW:
Groups:
- Imlifidase: Participants randomized to imlifidase
- Plasma Exchange: Participants randomized to plasma exchange
Period: Overall Study
Arm/Group | Imlifidase | Plasma Exchange
Started | 19 | 10
Completed | 17 | 10
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Imlifidase | Plasma Exchange | Total
Number analyzed (Participants) | 19 | 10 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (13.7) | 52.8 (16.4) | 46.8 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 11 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 0 | 5
  White | 14 | 9 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 1 | 3 | 4
  United States | 2 | 1 | 3
  France | 10 | 3 | 13
  Australia | 1 | 0 | 1
  Germany | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Maximum Reduction in Donor Specific Antibodies (DSA) Level During the 5 Days Following the Start of Treatment
Description: Maximum reduction (%) in the sum of DSA at any time point during the 5 days following the start of treatment.
  Only DSA with ≥1000 mean fluorescence intensity (MFI) at pre-treatment were included in the calculations.
  Clarification: The higher the maximum reduction percentage the lower the remaining DSA level.
Time Frame: Start of treatment until 5 days following start of treatment
Population: Participants with MFI values less than 1000 were excluded from the analysis
Measure: Mean (Standard Deviation); unit: percentage of maximum DSA reduction
Arm/Group | Imlifidase | Plasma Exchange
Number analyzed (Participants) | 18 | 8
percentage of maximum DSA reduction | 94 (4) | 36 (26)

2. Secondary Outcome: Reduction in DSA Levels After Treatment
Description: DSA levels were assessed at all visits throughout the study. The results are presented as reduction (%) from baseline. Clarification: The higher the reduction percentage the lower the remaining DSA level. Please observe that a negative reduction value represents an increase in DSA level from baseline.
Time Frame: Screening until Day 180
Measure: Mean (Standard Deviation); unit: percentage of DSA reduction
Arm/Group | Imlifidase | Plasma Exchange
Number analyzed (Participants) | 18 | 8
percentage of DSA reduction
  2 hours | 91 (7) | -2 (28)
  6 hours | 94 (4) | -2 (33)
  24 hours | 92 (5) | 0 (25)
  48 hours | 89 (10) | 18 (34)
  72 hours | 83 (24) | 10 (32)
  96 hours | 58 (32) | 22 (26)
  Day 6 | 41 (42) | 31 (23)
  Day 8 | 33 (45) | 39 (20)
  Day 11 | 35 (34) | 22 (34)
  Day 15 | 31 (43) | 28 (36)
  Day 22 | 28 (46) | 23 (34)
  Day 29 | 35 (30) | 30 (14)
  Day 64 | 30 (38) | 32 (34)
  Day 90 | 25 (41) | 41 (33)
  Day 180 | 29 (38) | 35 (32)

3. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR) Levels
Description: eGFR as calculated from p-creatinine is a measure of kidney function. eGFR was assessed at all visits throughout the study.
Time Frame: Screening until Day 180
Population: Some patients had missing values at sporadic occasions.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m2
Arm/Group | Imlifidase | Plasma Exchange
Number analyzed (Participants) | 19 | 10
mL/min/1.73m2
  Pre-dose: number analyzed (Participants) | 18 | 10
  Pre-dose | 28.0 (14.0) | 21.0 (8.1)
  24 hours | 25.8 (13.8) | 23.5 (11.0)
  48 hours | 26.2 (14.5) | 25.7 (9.4)
  72 hours | 27.6 (15.9) | 27.2 (10.8)
  96 hours | 30.6 (19.5) | 30.5 (13.8)
  Day 6: number analyzed (Participants) | 18 | 10
  Day 6 | 30.3 (18.6) | 31.2 (12.9)
  Day 8 | 33.4 (21.1) | 36.2 (18.2)
  Day 11: number analyzed (Participants) | 19 | 9
  Day 11 | 32.2 (18.9) | 34.0 (16.6)
  Day 15 | 32.1 (19.3) | 31.1 (15.4)
  Day 22 | 29.8 (16.7) | 31.9 (14.8)
  Day 29 | 27.5 (15.3) | 31.7 (14.5)
  Day 64: number analyzed (Participants) | 18 | 10
  Day 64 | 29.4 (14.9) | 34.6 (14.5)
  Day 90 | 27.2 (16.7) | 31.6 (12.8)
  Day 180: number analyzed (Participants) | 16 | 10
  Day 180 | 29.9 (15.5) | 32.5 (17.8)

4. Secondary Outcome: Urine Albumine/Creatinine Ratio
Description: The albumine/creatinine ratio in urine is a measure of kidney function.
Time Frame: Pre-dose until Day 180
Population: Some patients had missing data at different occasions during the study.
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Imlifidase | Plasma Exchange
Number analyzed (Participants) | 19 | 10
mg/g
  Pre-dose: number analyzed (Participants) | 16 | 9
  Pre-dose | 626 (972) | 134 (165)
  Day 90: number analyzed (Participants) | 18 | 9
  Day 90 | 669 (964) | 119 (166)
  Day 180: number analyzed (Participants) | 13 | 9
  Day 180 | 815 (1018) | 242 (295)

5. Secondary Outcome: Number of Patients With Graft Loss Within 180 Days of Treatment
Description: Information on patients who experienced graft loss was collected throughout the study.
Time Frame: Screening until Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Imlifidase | Plasma Exchange
Number analyzed (Participants) | 19 | 10
Participants | 5 | 0

6. Secondary Outcome: Number of Patients With Signs or no Signs of Transplant Glomerulopathy at Day 180
Description: Biopsies collected 180 days after treatment were analysed for signs of glomerulopathy.
Time Frame: Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Imlifidase | Plasma Exchange
Number analyzed (Participants) | 19 | 10
Participants
  Patients with no signs of transplant glomerulopathy | 7 | 4
  Patients with signs of transplant glomerulopathy | 8 | 6
  Patiens with no biopsy result or no evaluable biopsy result | 4 | 0

7. Secondary Outcome: Number of Patients With Different Types of Kidney Histopathology Throughout the Trial
Description: Kidney biopsies were assessed according to the Banff (2017) criteria at screening (baseline), Day 29, and Day 180.
  Abbreviations: AMR=Antibody mediated rejection, CMR=cell-mediated rejection
Time Frame: Screening, Day 29 and Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Imlifidase | Plasma Exchange
Number analyzed (Participants) | 19 | 10
Participants
  Screening: Active AMR | 7 | 4
  Screening: Active AMR + Borderline CMR | 0 | 1
  Screening: Active AMR + CMR | 5 | 1
  Screening: Chronic Active AMR + Borderline CMR | 3 | 1
  Screening: Chronic Active AMR + CMR | 1 | 2
  Screening: Chronic Active AMR | 3 | 1
  Screening: Borderline CMR | 0 | 0
  Screening: CMR | 0 | 0
  Screening: No rejection | 0 | 0
  Screening: Missing data | 0 | 0
  Day 29: Active AMR | 4 | 3
  Day 29: Active AMR + Borderline CMR | 0 | 1
  Day 29: Active AMR + CMR | 1 | 1
  Day 29: Chronic Active AMR + Borderline CMR | 1 | 1
  Day 29: Chronic Active AMR + CMR | 1 | 0
  Day 29: Chronic Active AMR | 4 | 2
  Day 29: Borderline CMR | 0 | 1
  Day 29: CMR | 1 | 0
  Day 29: No rejection | 5 | 1
  Day 29: Missing data | 2 | 0
  Day 180: Active AMR | 2 | 2
  Day 180: Active AMR + Borderline CMR | 0 | 0
  Day 180: Active AMR + CMR | 1 | 0
  Day 180: Chronic Active AMR + Borderline CMR | 2 | 0
  Day 180: Chronic Active AMR + CMR | 1 | 0
  Day 180: Chronic Active AMR | 5 | 5
  Day 180: Borderline CMR | 0 | 0
  Day 180: CMR | 0 | 1
  Day 180: No rejection | 2 | 2
  Day 180: Missing data | 6 | 0

8. Secondary Outcome: Number of Patients With Resolved AMR as Assessed by Messenger Ribonucleic Acid (mRNA) Levels
Description: Kidney biopsies were taken at screening, Day 29, and Day 180. Changes from baseline in mRNA levels were assessed as evidence of resolved AMR.
Time Frame: Screening, Day 29, and Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Imlifidase | Plasma Exchange
Number analyzed (Participants) | 19 | 10
Participants
  Day 29 | 0 | 0
  Day 180 | 0 | 0

9. Secondary Outcome: Number of Administered Plasma Exchange (PE) and Immunoadsorption (IA) Sessions
Description: Total number of administered PE and IA sessions to each treatment group are presented during the complete trial (Day 1 to Day 180) and for the time period: start of IVIg administration to Day 180.
Time Frame: Day 1 to Day 180
Population: In total 4 patients from the imlifidase arm were treated with PE. Of these 3 patients received PE after start of IVIg.
  All 10 patients from the PE arm were treated with PE. Of these 1 patient received PE after start of IVIg.
  One (1) patient from the PE arm also received IA after start of IVIg.
Measure: Number; unit: Sessions
Arm/Group | Imlifidase | Plasma Exchange
Number analyzed (Participants) | 19 | 10
Sessions
  Number of PE administered from Day 1 to Day 180: number analyzed (Participants) | 4 | 10
  Number of PE administered from Day 1 to Day 180 | 20 | 70
  Number of PE administered after start of IVIg: number analyzed (Participants) | 3 | 1
  Number of PE administered after start of IVIg | 18 | 11
  Number of IA administered from Day 1 to Day 180: number analyzed (Participants) | 19 | 1
  Number of IA administered from Day 1 to Day 180 | 0 | 23
  Number of IA administered after start of IVIg: number analyzed (Participants) | 19 | 1
  Number of IA administered after start of IVIg | 0 | 23

10. Secondary Outcome: Total Serum Immunoglobulin G (IgG) Levels Until Administration of Intravenous Immunoglobulin (IVIg)
Description: Total serum IgG levels over time following treatment until administration of IVIg.
  Please observe, IVIg was initiated on Day 4 (before 96 h measurement) for the imlifidase group.
Time Frame: Pre-dose until Day 6
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Imlifidase | Plasma Exchange
Number analyzed (Participants) | 19 | 10
mg/mL
  Pre-dose | 8.6 (6.1) | 7.9 (5.5)
  2 hours | 0.2 (0.1) | 4.3 (3.5)
  6 hours | 0.2 (0.1) | 4.6 (3.6)
  24 hours | 0.2 (0.2) | 5.2 (3.7)
  48 hours | 0.2 (0.2) | 4.6 (4.3)
  72 hours | 0.5 (0.8) | 4.8 (4.3)
  96 hours | 11.7 (5.4) | 4.1 (4.3)
  Day 6 | 20.0 (8.4) | 4.2 (4.5)

11. Secondary Outcome: Number of Patients With Intact IgG, Single-cleaved IgG (scIgG), F(ab')2 Fragments Following Treatment Until Administration of IVIg
Description: Presence of IgG, scIgG, and F(ab')2 was analysed using sodium dodecyl-sulphate polyacrylamide gel electrophoresis (SDS-PAGE)/western blot.
  Of note, IVIg was administered on Day 4 (before 96 h measurement) to patients treated with imlifidase. Hence no analyses beyond this timepoint were performed for this group.
Time Frame: Start of treatment (Day 1) up to administration of IVIg on Day 4 (imlifidase group) and until administration of IVIg within Day 15 (PE group)
Population: IVIg was administered on Day 4 (before 96 h measurement) to patients treated with imlifidase. Hence measurement of intact IgG was not performed for this group from 96 hours onwards. Measurement was stopped for PE patients when IVIg was administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Imlifidase | Plasma Exchange
Number analyzed (Participants) | 19 | 10
Participants
  Baseline: Only intact IgG | 19 | 10
  Baseline: Mix of intact IgG and scIgG | 0 | 0
  Baseline: Only scIgG | 0 | 0
  Baseline: Mix of scIgG and F(ab')2 | 0 | 0
  Baseline: Only F(ab')2 | 0 | 0
  Baseline: No intact IgG, scIgG, or F(ab')2 | 0 | 0
  2 hours: Only intact IgG | 0 | 10
  2 hours: Mix of intact IgG and scIgG | 0 | 0
  2 hours: Only scIgG | 0 | 0
  2 hours: Mix of scIgG and F(ab')2 | 2 | 0
  2 hours: Only F(ab')2 | 17 | 0
  2 hours: No intact IgG, scIgG, or F(ab')2 | 0 | 0
  6 hours: Only intact IgG | 0 | 10
  6 hours: Mix of intact IgG and scIgG | 0 | 0
  6 hours: Only scIgG | 0 | 0
  6 hours: Mix of scIgG and F(ab')2 | 0 | 0
  6 hours: Only F(ab')2 | 19 | 0
  6 hours: No intact IgG, scIgG, or F(ab')2 | 0 | 0
  24 hours: Only intact IgG | 0 | 9
  24 hours: Mix of intact IgG and scIgG | 0 | 0
  24 hours: Only scIgG | 0 | 0
  24 hours: Mix of scIgG and F(ab')2 | 0 | 0
  24 hours: Only F(ab')2 | 19 | 0
  24 hours: No intact IgG, scIgG, or F(ab')2 | 0 | 1
  48 hours: Only intact IgG | 0 | 8
  48 hours: Mix of intact IgG and scIgG | 0 | 0
  48 hours: Only scIgG | 0 | 0
  48 hours: Mix of scIgG and F(ab')2 | 1 | 0
  48 hours: Only F(ab')2 | 18 | 0
  48 hours: No intact IgG, scIgG, or F(ab')2 | 0 | 2
  72 hours: Only intact IgG | 0 | 10
  72 hours: Mix of intact IgG and scIgG | 2 | 0
  72 hours: Only scIgG | 0 | 0
  72 hours: Mix of scIgG and F(ab')2 | 1 | 0
  72 hours: Only F(ab')2 | 16 | 0
  72 hours: No intact IgG, scIgG, or F(ab')2 | 0 | 0
  96 hours: number analyzed (Participants) | 0 | 10
  96 hours: Only intact IgG | 0 | 9
  96 hours: Mix of intact IgG and scIgG | 0 | 0
  96 hours: Only scIgG | 0 | 0
  96 hours: Mix of scIgG and F(ab')2 | 0 | 0
  96 hours: Only F(ab')2 | 0 | 0
  96 hours: No intact IgG, scIgG, or F(ab')2 | 0 | 1
  Day 6: number analyzed (Participants) | 0 | 10
  Day 6: Only intact IgG | 0 | 10
  Day 6: Mix of intact IgG and scIgG | 0 | 0
  Day 6: Only scIgG | 0 | 0
  Day 6: Mix of scIgG and F(ab')2 | 0 | 0
  Day 6: Only F(ab')2 | 0 | 0
  Day 6: No intact IgG, scIgG, or F(ab')2 | 0 | 0
  Day 8: number analyzed (Participants) | 0 | 8
  Day 8: Only intact IgG | 0 | 8
  Day 8: Mix of intact IgG and scIgG | 0 | 0
  Day 8: Only scIgG | 0 | 0
  Day 8: Mix of scIgG and F(ab')2 | 0 | 0
  Day 8: Only F(ab')2 | 0 | 0
  Day 8: No intact IgG, scIgG, or F(ab')2 | 0 | 0
  Day 11: number analyzed (Participants) | 0 | 5
  Day 11: Only intact IgG | 0 | 5
  Day 11: Mix of intact IgG and scIgG | 0 | 0
  Day 11: Only scIgG | 0 | 0
  Day 11: Mix of scIgG and F(ab')2 | 0 | 0
  Day 11: Only F(ab')2 | 0 | 0
  Day 11: No intact IgG, scIgG, or F(ab')2 | 0 | 0
  Day 15: number analyzed (Participants) | 0 | 2
  Day 15: Only intact IgG | 0 | 1
  Day 15: Mix of intact IgG and scIgG | 0 | 0
  Day 15: Only scIgG | 0 | 0
  Day 15: Mix of scIgG and F(ab')2 | 0 | 0
  Day 15: Only F(ab')2 | 0 | 0
  Day 15: No intact IgG, scIgG, or F(ab')2 | 0 | 1

12. Secondary Outcome: DSA Functionality Determined by C1q Analysis Pre- and Post-treatment
Description: An MFI value above 6000 is indicative of complement fixation. Analysis of DSA functionality assessed as mean MFI levels was done before and after treatment.
Time Frame: Screening until Day 6
Population: Data was missing for a number of patients.
Measure: Mean (Standard Deviation); unit: MFI counts
Arm/Group | Imlifidase | Plasma Exchange
Number analyzed (Participants) | 19 | 10
MFI counts
  Pre-dose: number analyzed (Participants) | 11 | 6
  Pre-dose | 19827 (11910) | 18848 (9958)
  Day 2: number analyzed (Participants) | 11 | 6
  Day 2 | 319 (432) | 15576 (12008)
  Day 6: number analyzed (Participants) | 10 | 6
  Day 6 | 5065 (9768) | 11926 (13076)

13. Secondary Outcome: Pharmacokinetic (PK) Profile of Imlifidase: Cmax
Description: Cmax = Maximum observed plasma concentration of imlifidase following dosing
Time Frame: Pre-dose, 30 min, 1 h, 2 h, 6 h, 24 h, 48 h, 72 h, 96 h, Day 6, Day 8, Day 1, and Day 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- PK Analysis Set: Patients treated with imlifidase
Arm/Group | PK Analysis Set
Number analyzed (Participants) | 19
µg/mL | 4.3 (18)

14. Secondary Outcome: PK Profile of Imlifidase: Tmax
Description: Tmax = Time point for maximum observed plasma concentration of imlifidase following dosing
Time Frame: Pre-dose, 30 min, 1 h, 2 h, 6 h, 24 h, 48 h, 72 h, 96 h, Day 6, Day 8, Day 1, and Day 15
Measure: Median (Full Range); unit: h
Arm/Group | PK Analysis Set
Number analyzed (Participants) | 19
h | 0.6 [0.4 to 2.3]

15. Secondary Outcome: PK Profile of Imlifidase: t1/2
Description: t1/2 = terminal half-life of imlifidase (refers to the time required for plasma concentration of a drug to decrease by 50%) Different mathematical models are available to describe how drugs are adsorbed, distributed, metabolised, and eliminated from the body. The time-concentration curve of imlifidase could be fitted to the so called 2-compartment model. This model divide the body into a central and an peripheral compartment. The central compartment consist of the plasma and tissues where the distribution is fast and the peripheral consists of tissues where the distribution of the drug is slower. As a result the elimination of imlifidase consists of an initial phase with a short half life (alpha-t1/2) and an elimination phase with a longer half-life (beta-t1/2).
Time Frame: Pre-dose, 30 min, 1 h, 2 h, 6 h, 24 h, 48 h, 72 h, 96 h, Day 6, Day 8, Day 1, and Day 15
Population: The data presents only patients who's time-concentration profile could be fitted to a 2-compartment model
Measure: Median (Full Range); unit: h
Arm/Group | PK Analysis Set
Number analyzed (Participants) | 19
h
  Alpha t1/2 (initial phase) | 2.7 [1.4 to 6.0]
  Beta t1/2 (elimination phase): number analyzed (Participants) | 16
  Beta t1/2 (elimination phase) | 39.7 [23.5 to 128.0]

16. Secondary Outcome: PK Profile of Imlifidase: AUC
Description: Area under the imlifidase plasma concentration vs time curve (AUC)
Time Frame: Pre-dose, 30 min, 1 h, 2 h, 6 h, 24 h, 48 h, 72 h, 96 h, Day 6, Day 8, Day 1, and Day 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h×µg/mL
Arm/Group | PK Analysis Set
Number analyzed (Participants) | 16
h×µg/mL | 124 (62)

17. Secondary Outcome: PK Profile of Imlifidase: CL
Description: Clearance (CL) of imlifidase means the volume of blood cleared of imlifidase per unit of time.
Time Frame: Pre-dose, 30 min, 1 h, 2 h, 6 h, 24 h, 48 h, 72 h, 96 h, Day 6, Day 8, Day 1, and Day 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h/kg
Arm/Group | PK Analysis Set
Number analyzed (Participants) | 16
mL/h/kg | 2.0 (62)

18. Secondary Outcome: PK Profile of Imlifidase: Volume of Distribution (V)
Description: Vss = volume of distribution associated with steady state VZ = volume of distribution associated with the elimination phase
Time Frame: Pre-dose, 30 min, 1 h, 2 h, 6 h, 24 h, 48 h, 72 h, 96 h, Day 6, Day 8, Day 1, and Day 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/kg
Arm/Group | PK Analysis Set
Number analyzed (Participants) | 16
L/kg
  Vss | 0.64 (722)
  Vz | 0.54 (547)

19. Secondary Outcome: Concentration of Anti-drug Antibodies (ADAs)
Description: Samples were collected and analysed for presence of anti-imlifidase IgG throughout the study.
  Imlifidase is an IgG-degrading enzyme of Streptococcus pyogenes. Patients who have been exposed to Streptococcus prior to participating in this trial tested positive for ADA also before exposure to imlifidase.
Time Frame: Screening until Day 180
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | PK Analysis Set
Number analyzed (Participants) | 19
mg/L
  Pre-dose | 6.7 (70)
  24 hours | 2.0 (0)
  Day 8 | 15 (66)
  Day 11 | 20 (149)
  Day 15 | 49 (275)
  Day 22 | 73 (300)
  Day 29 | 87 (398)
  Day 64 | 122 (496)
  Day 90 | 135 (536)
  Day 180 | 100 (725)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for 6 months (i.e., from the timepoint the participant signed the informed consent form (ICF) until end of study, including the follow-up period). AEs occurring after the start of trial treatment and within the time of residual drug effect which is 28 days after start of trial treatment are classified as treatment emergent AEs (TEAEs).
Description: AEs were obtained if spontaneously reported, if reported in response to an open question from the study personnel or if revealed by observation.
  The reported data consists of TEAEs regardless of whether they are considered treatment-related or non-treatment-related.
  The reported data on mortality includes the 6 months follow-up period.
Arm/Group | Imlifidase | Plasma Exchange
All-Cause Mortality (participants affected / at risk) | 1/19 | 0/10
Serious Adverse Events (participants affected / at risk) | 3/19 | 3/10
Other Adverse Events (participants affected / at risk) | 17/19 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imlifidase (N=19) | Plasma Exchange (N=10)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imlifidase (N=19) | Plasma Exchange (N=10)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (5) | 1 (1)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 3 (3) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Transplant rejection (Immune system disorders) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Renal lymphocele (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acid base balance abnormal (Investigations) | 1 (1) | 0 (0)
Antibody test positive (Investigations) | 1 (1) | 0 (0)
BK polyomavirus test positive (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 3 (3) | 1 (3)
Blood glucose fluctuation (Investigations) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 2 (2) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 2 (2)
Immunosuppressant drug level increased (Investigations) | 1 (1) | 0 (0)
Calcium deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (10) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (4) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Feeling of despair (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the study, one or more manuscripts for joint publication may be prepared in collaboration between the investigator(s) offered authorship and Hansa Biopharma.

Any confidential information relating to imlifidase or the study, including any data and results from the study will be the exclusive property of Hansa Biopharma AB. The investigators and any other persons involved in the trial will protect the confidentiality of the proprietary information belonging to Hansa Biopharma AB.

DOCUMENTS (2):
  • Study Protocol (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/05/NCT03897205/Prot_001.pdf
  • Statistical Analysis Plan (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT03897205/SAP_002.pdf